CLINICAL TRIAL: NCT05442398
Title: Detection of Celiac Disease Among Suspected Patients With Type 1 Diabetes Mellitus
Brief Title: Celiac Disease and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Mohamed Salah Ahmed Ali (Other)
Responsible Party: Sponsor-Investigator, Mohamed Salah Ahmed Ali, Physician, Assiut University
Organization: Assiut University (Other)
Other Study IDs: celiac and diabetes
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Celiac Disease in Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to detect Celiac Disease among suspected patients with Type 1 Diabetes Mellitus who admitted to Assiut University Children's Hospital during one year duration

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is an immune-mediated disease characterized by reduced insulin secretion by islet Beta cells in the pancreas that leads to insulin deficiency . Because of a common genetic background and interaction between environmental and immunological factors, Patients with T1DM are at a great risk for developing autoimmune diseases. It is well recognized that T1DM can be associated with celiac disease (CD) and autoimmune thyroid disorders (ATD). Recent studies regarding CD and T1DM have indicated that the frequency of this association can vary from 1.7% to 16% . Also other autoimmune diseases may be noted such as Addison's disease and vitiligo.

Celiac disease is an autoimmune enteropathy that is caused by permanent susceptibility to gluten (a protein found in wheat, barley, and rye) in genetically susceptible individuals .

CD develops with symptoms, such as steatorrhea, weight loss, developmental disorder, abdominal pain, and nutritional symptoms (e.g. vitamin deficiency), and is improved shortly after elimination of gluten-containing foods .

Extraintestinal signs and symptoms include iron-deficiency anemia, chronic fatigue, failure to thrive, stunted or short stature, delayed puberty, amenorrhea, recurrent aphthous stomatitis, dermatitis herpetiformis - like rash, fracture with inadequate traumas, osteopenia, osteoporosis.

Since the majority of CD patients can be asymptomatic, screening for CD at the time of T1DM diagnosis is recommended . In seronegative cases at the first screening, if there are no CD symptoms, regular screening every 2-5 years is recommended. However, in patients with CD symptoms or history of CD in first-degree relatives more frequent screening is recommended . Testing of asymptomatic CD would provide a prompt diagnosis of CD and enable better metabolic control for T1DM patients .

However, recently, some studies have shown normalization of celiac serology in patients with T1DM, even with no gluten-free dietary intervention. In the mentioned studies, spontaneous normalization developed in 20-35% of the cases

. Therefore, considering all of the serologically positive individuals as CD and giving a gluten-free diet (GFD) imposes an additional psychological burden for children and families.

In the latest European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) guidelines, it was highlighted that the level of anti-tissue transglutaminase-IgA (anti-TTG IgA) should be at least 10 times higher than the upper limit of normal (ULN) for diagnosis of CD without duodenal biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes mellitus
* Symptoms and signs suggestive of Celiac disease.
* Age : 1-18 years old

Exclusion Criteria:

* No symptoms or signs suggestive of celiac disease.
* Patients who are Non CD gluten hypersensitivity
* Age : less than 1 year old.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sample size was calculated using Epi- Info7. There was no previous studies that calculate the percentage of Children from 1-18 years old diagnosed as Type 1 Diabetes mellitus with Symptoms and signs suggestive of Celiac disease, we hypothesized that the percentage will be 50% . Based on this percentage and with a confidence limits of 10% and a confidence level of 80%, the minimum sample needed for the study was estimated to be 41 patients.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Anti-tissue transglutaminase (anti-tTG) antibodies IgA-IgG | within 2 weeks
  negative less than 10 positive if more than 10
Total IGA | within 2 weeks
  normal range 61-348
HbA1c | 1 day visit
  Less than 5.7% Pre-diabetes: 5.7% to 6.4% Diabetes: 6.5% or higher

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Tawfeek, Professor, Study Chair — Assiut University
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volta U, Tovoli F, Caio G. Clinical and immunological features of celiac disease in patients with Type 1 diabetes mellitus. Expert Rev Gastroenterol Hepatol. 2011 Aug;5(4):479-87. doi: 10.1586/egh.11.38. PMID 21780895
- [Background] Scaramuzza AE, Mantegazza C, Bosetti A, Zuccotti GV. Type 1 diabetes and celiac disease: The effects of gluten free diet on metabolic control. World J Diabetes. 2013 Aug 15;4(4):130-4. doi: 10.4239/wjd.v4.i4.130. PMID 23961323
- [Background] Husby S, Koletzko S, Korponay-Szabo I, Kurppa K, Mearin ML, Ribes-Koninckx C, Shamir R, Troncone R, Auricchio R, Castillejo G, Christensen R, Dolinsek J, Gillett P, Hrobjartsson A, Koltai T, Maki M, Nielsen SM, Popp A, Stordal K, Werkstetter K, Wessels M. European Society Paediatric Gastroenterology, Hepatology and Nutrition Guidelines for Diagnosing Coeliac Disease 2020. J Pediatr Gastroenterol Nutr. 2020 Jan;70(1):141-156. doi: 10.1097/MPG.0000000000002497. PMID 31568151
- [Background] Fasano A, Catassi C. Clinical practice. Celiac disease. N Engl J Med. 2012 Dec 20;367(25):2419-26. doi: 10.1056/NEJMcp1113994. No abstract available. PMID 23252527
- [Background] Green PH, Cellier C. Celiac disease. N Engl J Med. 2007 Oct 25;357(17):1731-43. doi: 10.1056/NEJMra071600. No abstract available. PMID 17960014
- [Background] Chiang JL, Maahs DM, Garvey KC, Hood KK, Laffel LM, Weinzimer SA, Wolfsdorf JI, Schatz D. Type 1 Diabetes in Children and Adolescents: A Position Statement by the American Diabetes Association. Diabetes Care. 2018 Sep;41(9):2026-2044. doi: 10.2337/dci18-0023. Epub 2018 Aug 9. No abstract available. PMID 30093549
- [Background] Jabri B, Kasarda DD, Green PH. Innate and adaptive immunity: the yin and yang of celiac disease. Immunol Rev. 2005 Aug;206:219-31. doi: 10.1111/j.0105-2896.2005.00294.x. PMID 16048552
- [Background] Mahmud FH, Elbarbary NS, Frohlich-Reiterer E, Holl RW, Kordonouri O, Knip M, Simmons K, Craig ME. ISPAD Clinical Practice Consensus Guidelines 2018: Other complications and associated conditions in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2018 Oct;19 Suppl 27(Suppl 27):275-286. doi: 10.1111/pedi.12740. No abstract available. PMID 30066458
- [Background] Iughetti L, Bulgarelli S, Forese S, Lorini R, Balli F, Bernasconi S. Endocrine aspects of coeliac disease. J Pediatr Endocrinol Metab. 2003 Jul-Aug;16(6):805-18. doi: 10.1515/jpem.2003.16.6.805. PMID 12948292
- [Background] Ergur AT, Ocal G, Berberoglu M, Adiyaman P, Siklar Z, Aycan Z, Evliyaoglu O, Kansu A, Girgin N, Ensari A. Celiac disease and autoimmune thyroid disease in children with type 1 diabetes mellitus: clinical and HLA-genotyping results. J Clin Res Pediatr Endocrinol. 2010;2(4):151-4. doi: 10.4274/jcrpe.v2i4.151. Epub 2010 Nov 3. PMID 21274314
- [Background] Odeh R, Alassaf A, Gharaibeh L, Ibrahim S, Khdair Ahmad F, Ajlouni K. Prevalence of celiac disease and celiac-related antibody status in pediatric patients with type 1 diabetes in Jordan. Endocr Connect. 2019 Jun 13;8(6):780-787. doi: 10.1530/EC-19-0146. PMID 31085767
- [Background] Unal E, Demiral M, Baysal B, Agin M, Devecioglu EG, Demirbilek H, Ozbek MN. Frequency of Celiac Disease and Spontaneous Normalization Rate of Celiac Serology in Children and Adolescent Patients with Type 1 Diabetes. J Clin Res Pediatr Endocrinol. 2021 Feb 26;13(1):72-79. doi: 10.4274/jcrpe.galenos.2020.2020.0108. Epub 2020 Aug 21. PMID 32820875